CLINICAL TRIAL: NCT04507490
Title: Acute Effect of Whole Body Vibration of Different Frequencies on Balance and Functional Mobility of Patients With Parkinson: Crossover-type Controlled Clinical Trial
Brief Title: Analysis of Balance and Mobility for Parkinson Disease After Whole Body Vibration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, Maria das Graças Rodrigues de Araújo, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Whole_body_vibration_PD
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Balance; Function Mobility; Whole body vibration
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: After confirming the eligibility criteria, patients will be asked to sign the informed consent form. Subsequently, they will be randomly allocated to three groups: (i) group 6 Hz: full body vibration (frequency 6 Hz, amplitude 4 mm, five cycles lasting 1 minutes and interval between cycles of 1 minute) , (ii) 25 Hz group: full body vibration (25 Hz frequency, 4 mm amplitude, five cycles lasting 1 minute and interval between 1 minute cycles) and (iii) sham group: The sham vibration will be performed with the platform disconnected. Additionally, a sound device will be connected producing a noise similar to that of the connected platform for a time equivalent to that of the treatment protocol. The patient will be instructed to position himself standing on the platform, with a semi knee flexion in order that the vibration wave does not propagate to the head. There will be a washout time of at least one week between one intervention and another
Who Masked: Participant, Investigator
Masking Description: Double blind. Only the interventionist will be allowed to access the vibration condition. In this way, the patient and the investigator will be blind for the type of vibration that the patient will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole body vibration 6 Hz (Experimental): application of whole body vibration in the following parameters:frequency 6 Hz, amplitude 4 mm, five cycles lasting 1 minutes and interval between cycles of 1 minute
  Interventions: Device: Whole body vibration
- Whole body vibration 25 Hz (Experimental): application of whole body vibration in the following parameters: 25 Hz frequency, 4 mm amplitude, five cycles lasting 1 minute and interval between 1 minute cycles
  Interventions: Device: Whole body vibration
- Whole body vibration sham (Sham Comparator): application of whole body vibration in the following parameters: The sham vibration will be performed with the platform disconnected. A sound device will be connected producing a noise similar to that of the connected platform for a time equivalent to that of the treatment protocol.
  Interventions: Device: Whole body vibration

INTERVENTIONS:
Device: Whole body vibration — 315/5000 application of whole body vibration with pre-established parameters for each group. All patients will participate in all groups, an interval of at least one week. They will be instructed to climb on the platform and to position a semi knee flexion and remain stationary during the vibration

SUMMARY:
Parkinson's disease has innumerous motor symptoms that impacting on the functional level of the patient, such as impairment in functional mobility and balance . Previous studies have already aimed to evaluate the effectiveness of whole body vibration, but without methodological criteria. The use of whole body vibration may be an alternative for the treatment of Parkinson's disease. Therefore, the objective of the study is to verify which frequency of vibration is able to improve the balance and mobility of patients with Parkinson's disease.

DETAILED DESCRIPTION:
After confirming the eligibility criteria, patients will be asked to sign the informed consent form. Subsequently, they will be randomly allocated to three groups: (i) group 6 Hz: full body vibration (frequency 6 Hz, amplitude 4 mm, five cycles lasting 1 minutes and interval between cycles of 1 minute) , (ii) 25 Hz group: full body vibration (25 Hz frequency, 4 mm amplitude, five cycles lasting 1 minute and interval between 1 minute cycles) and (iii) sham group: The sham vibration will be performed with the platform disconnected. Additionally, a sound device will be connected producing a noise similar to that of the connected platform for a time equivalent to that of the treatment protocol. The patient will be instructed to position himself standing on the platform, with a semi knee flexion in order that the vibration wave does not propagate to the head. The allocation will be made randomly among individuals, using a random sequence table generated by the website www.randomization.com. There will be a washout time of at least one week between one intervention and another. All evaluations took place inside the laboratory, which has all the equipment for the evaluation. The evaluations will take place immediately before the intervention and immediately after.

ELIGIBILITY:
Inclusion Criteria:

* · Minimum score of the Montreal Cognitive Assessment (MoCA) (27 points);

  * Regular antiparkinsonian pharmacological treatment;
  * Staged from I to III on the modified Hoehn & Yahr scale.

Exclusion Criteria:

* · Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests;

  * other associated neurological disease
  * changes in medication in use for Parkinson's disease for at least sixty days before the start of the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Function mobility | Before (T0) and immediate after vibration (T1)
  The evaluation of the functional mobility of individuals will be performed by the Timed Up and Go test. It will analyze the time spent by the individual to get up from a chair with arms, walk for three meters and return to the chair
Change in Static and dynamic balance | Before (T0) and immediate after vibration (T1)
  The assessment of static and dynamic balance using the Biodex Balance System (BBS) tool, capable of evaluating the displacement of the center of mass in the anteroposterior and laterolateral axes on a circular platform that can oscillate up to 20 ° in all directions in the horizontal plane. Static balance was performed using the Postural Stability Test, while dynamic balance was assessed using the Limits of Stability Test. The MiniBest test was performed to assess dynamic balance. The test consists of the application of 14 tasks that measure the patient's dynamic balance in different positions, through 14 items, with scores ranging from zero to two
Change in static balance | Before (T0) and immediate after vibration (T1)
  The indirect center of pressure (COP) was acquired by the baropodometric static platform (Sensor Medica). The patient was instructed to position himself on the platform with his arms relaxed along his body, in the usual posture and looking towards the horizon, with a postural adaptation time of 30 seconds. The collection started without being informed to the patient. The averages of the three acquisitions of the following measures were analyzed of center of pressure
Change in foot pressure | Before (T0) and immediate after vibration (T1)
  The direct foot pressure was acquired by the baropodometric static platform (Sensor Medica).The patient was instructed to position himself on the platform with his arms relaxed along his body, in the usual posture and looking towards the horizon, with a postural adaptation time of 30 seconds. The collection started without being informed to the patient. The averages of the three acquisitions of the following measures were analyzed: (i) maximum pressure in the forefoot; (ii) maximum pressure in the midfoot and (iii) maximum pressure in the hindfoot.

SECONDARY OUTCOMES:
Change in Cadence of gait | Before (T0) and immediate after vibration (T1)
  The acquisition was made during the timed up and go, using the Wiva® Mob, an inertial sensor connected to the software via Bluetooth. The inertial sensor will be placed on the patient's waist to measure gait cadence during the timed up ando go test
Change in support phase of gait | Before (T0) and immediate after vibration (T1)
  The acquisition was made during the timed up and go, using the Wiva® Mob, an inertial sensor connected to the software via Bluetooth. The inertial sensor will be placed on the patient's waist to measure gait support phase during the timed up ando go test
Change in swing phase of gait | Before (T0) and immediate after vibration (T1)
  The acquisition was made during the timed up and go, using the Wiva® Mob, an inertial sensor connected to the software via Bluetooth. The inertial sensor will be placed on the patient's waist to measure gait swing phase during the timed up ando go test
Change in Risk of falls | Before (T0) and immediate after vibration (T1)
  It was assessed using the "FallRisk" test of the Biodex balance System balance platform. The BBS will show the general stability index (GSI). In addition to the GSI, the BBS will show whether the patient is at risk of falls considering the age group
Change in Functionality assessment | Before (T0) and immediate after vibration (T1)
  It was carried out through session III of the UPDRS (Unified parkinson's disease rating scale), the responses vary between 0 and 4 with a total sum of the items of 108, so that higher values indicate a greater degree of dependence, while, lower values, greater degree of functionality

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Mendes, Paulista, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No